CLINICAL TRIAL: NCT01275937
Title: A Double Blind Study Comparing Low Dose and High Dose IV Esomeprazole After Successful Endoscopic Therapy in Patients With Peptic Ulcer Bleeding
Brief Title: A Double Blind Study Comparing Two Doses of IV Esomeprazole After Successful Endoscopic Therapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University (Other)
Responsible Party: Lin Hwai-Jeng, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TMUH-2011
Record Dates: First submitted 2011-01-12; First posted 2011-01-13 (Estimated); Last update posted 2011-08-12 (Estimated); Status verified 2011-08

CONDITIONS: Upper Gastrointestinal Bleeding
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Esomeprazole (Other): Esomeprazole 40 mg IV daily is given for three days followed by40mg once daily orally for two months.
  Interventions: Drug: Esomeprazole
- esomeprazole (Active Comparator): esomeprazole 160 mg/day continuous infusion is given for three days followed by 40mg once daily orally for two months.
  Interventions: Drug: Esomeprazole

INTERVENTIONS:
Drug: Esomeprazole — Esomeprazole 40 mg IV daily is given for three days. Thereafter, the patients receive 40 mg Esomeprazole orally daily for two months.
Drug: esomeprazole — esomeprazole 160 mg/day continuous infusion is given for three days. Thereafter, the patients receive 40 mg nexium orally daily for two months.
  Other Names: nexium

SUMMARY:
A bleeding peptic ulcer remains a serious medical problem with significant morbidity and mortality. Endoscopic therapy significantly reduces further bleeding, surgery, and mortality in patients with bleeding peptic ulcers and is now recommended as the first hemostatic modality for these patients.

In the past few years, adjuvant use of a high-dose proton pump inhibitor (PPI) after endoscopic therapy has been endorsed in some studies. However, low dose of PPI has also been supported in the management of these patients.

The investigators enroll 130 patients with active bleeding or nonbleeding visible vessels in this study. They are randomly assigned as 40 mg/day or 160mg/day IV nexium group. All patients receive successful endoscopic therapy with heater probe or hemoclip placement.

In the low dose group (N=65), 40 mg IV Nexium daily is given for three days. Thereafter, the patients receive 40 mg nexium orally daily for two months. In the large dose group (N=65), 160 mg/day continuous infusion is given for three days. Thereafter, the patients receive 40 mg nexium orally daily for two months.

The primary end point is recurrent bleeding before discharge and within 14 days. At day 14, volume of blood transfused, number of surgeries performed, and the mortality rates of the two groups are compared as well.

DETAILED DESCRIPTION:
A bleeding peptic ulcer remains a serious medical problem with significant morbidity and mortality. Endoscopic therapy significantly reduces further bleeding, surgery, and mortality in patients with bleeding peptic ulcers and is now recommended as the first hemostatic modality for these patients.

In the past few years, adjuvant use of a high-dose proton pump inhibitor (PPI) after endoscopic therapy has been endorsed in some studies. However, low dose of PPI has also been supported in the management of these patients.

We enroll 130 patients with active bleeding or nonbleeding visible vessels in this study. They are randomly assigned as 40 mg/day or 160mg/day IV nexium group. All patients receive successful endoscopic therapy with heater probe or hemoclip placement.

In the low dose group (N=65), 40 mg IV Nexium daily is given for three days. Thereafter, the patients receive 40 mg nexium orally daily for two months. In the large dose group (N=65), 160 mg/day continuous infusion is given for three days. Thereafter, the patients receive 40 mg nexium orally daily for two months.

The primary end point is recurrent bleeding before discharge and within 14 days. At day 14, volume of blood transfused, number of surgeries performed, and the mortality rates of the two groups are compared as well.

ELIGIBILITY:
Inclusion Criteria:

* a peptic with active bleeding, a non-bleeding visible vessel or an adherent blood clot at the ulcer base is observed within24 hours of hospital admission

Exclusion Criteria:

* Patients are excluded from the study if they are pregnant, do not obtain initial hemostasis with endoscopic injection epinephrine, do not give written informed consent,have bleeding tendency(platelet count <50*109/L,serum prothrombin <30% of normal, or were taking anticoagulants), uremia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2011-08; Primary Completion 2013-12 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Two different doses intravenous proton pump inhibitors in patients with peptic ulcer bleeding after successful endoscopic therapy- a prospective randomized comparative trial. | two years
  recurrent bleeding before discharge and within 14 days

SECONDARY OUTCOMES:
Two different doses intravenous proton pump inhibitors in patients with peptic ulcer bleeding after successful endoscopic therapy- a prospective randomized comparative trial. | two years

CONTACTS AND LOCATIONS:
Overall Officials: Hwai-jeng Lin, MD, Study Chair — Taipei Medical University
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan, Taiwan